CLINICAL TRIAL: NCT05998590
Title: Pre-sleep Protein Supplementation Does Not Improve Performance, Body Composition and Recovery in British Army Recruits
Brief Title: Pre-sleep Protein Supplementation in British Army Recruits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1076/MODREC/20
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Protein-energy; Imbalance; Recovery; Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High protein intake supplementation (Experimental): A daily 60g dose of whey protein supplementation received between 8-9pm during BT.
  Interventions: Dietary Supplement: High protein supplement
- Moderate protein intake supplementation (Experimental): A daily 20g dose of whey protein supplementation received between 8-9pm during BT.
  Interventions: Dietary Supplement: Moderate protein supplement
- Carbohydrate placebo supplementation (Placebo Comparator): A daily isocaloric carbohydrate (maltodextrin) placebo received between 8-9pm during BT.
  Interventions: Dietary Supplement: Carbohydrate placebo
- Control group (Other): Control group, no daily supplement received, only participating in BT.
  Interventions: Other: Control: No supplementation

INTERVENTIONS:
Dietary Supplement: High protein supplement — The participants received a 60g protein bolus each evening prior to sleep from week 3 to week 12 of training.
  Arms: High protein intake supplementation
Dietary Supplement: Moderate protein supplement — The participants received a 20g protein bolus each evening prior to sleep from week 3 to week 12 of training.
  Arms: Moderate protein intake supplementation
Dietary Supplement: Carbohydrate placebo — The participants received an isocaloric carbohydrate bolus each evening prior to sleep from week 3 to week 12 of training.
  Arms: Carbohydrate placebo supplementation
Other: Control: No supplementation — The participants did not receive any supplementation but instead acted as a control group doing BT only
  Arms: Control group

SUMMARY:
Dietary protein has been shown to be important to support physical training. For occupational demands such as military training, new recruits often fail to meet the recommended protein intake during basic training (BT), with negligible amounts consumed in the evening. As such, individuals undertaking BT may require higher intakes than the general population.This study assessed the influence of a daily bolus of protein prior to sleep on performance adaptations, body composition and recovery in British Army recruits.

DETAILED DESCRIPTION:
Dietary protein is crucial for optimising physical training adaptations such as muscular strength and mass, which are key aims for athletic populations, including British Army recruits. New recruits fail to meet the recommended protein intake during basic training (BT), with negligible amounts consumed in the evening. This study aimed to assess the influence of a daily bolus of protein prior to sleep on performance adaptations, body composition and recovery in British Army recruits. The study will recruit a mixed cohort of >120 new recruits from the United Kingdom (UK) British Army who will be randomised into a dietary control (CON), carbohydrate placebo (PLA), moderate (20g) protein (MOD) or high (60g) protein (HIGH) supplementation group. Supplements will be isocaloric and consumed daily on weekday evenings between 2000 and 2100h for 10 weeks during BT, alongside standardised dietary intake and BT activities. Performance tests (mid-thigh pull, medicine ball throw, 2km run time, maximal push-up and maximal vertical jump) and body composition will be assessed at the start and end of BT under standardised conditions. Dietary intake, energy expenditure, salivary hormones, urinary nitrogen balance, perceived muscle soreness, rating of perceived exertion, mood and fatigue will be assessed at the start, middle and end of BT. The underlying aim of this study is to assess whether inclusion of nocturnal protein supplementation will influence performance adaptations, body composition changes or acute recovery in British Army recruits.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled into British Army basic training
* Medically fit to start Army training

Exclusion Criteria:

* Not taking any other nutritional supplement
* Not currently pregnant
* Not dairy or lactose intolerant or have any specific dietary requirements .

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Lower body strength performance | 12 weeks
  Mid-thigh pull

SECONDARY OUTCOMES:
Body composition | 12 weeks
  Fat-free mass

CONTACTS AND LOCATIONS:
Overall Officials: Justin D Roberts, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Anglia Ruskin University, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chapman S, Roberts J, Roberts AJ, Ogden H, Izard R, Smith L, Chichger H, Struszczak L, Rawcliffe AJ. Pre-sleep protein supplementation does not improve performance, body composition, and recovery in British Army recruits (part 1). Front Nutr. 2023 Nov 30;10:1262044. doi: 10.3389/fnut.2023.1262044. eCollection 2023. PMID 38144428